CLINICAL TRIAL: NCT00952588
Title: A Randomised, Open-label, Multi-centre, 2-stage, Parallel Group Study to Assess the Efficacy, Safety and Tolerability of AZD1152 Alone and in Combination With Low Dose Cytosine Arabinoside (LDAC) in Comparison With LDAC Alone in Patients Aged ≥ 60 With Newly Diagnosed Acute Myeloid Leukaemia (AML)
Brief Title: Study to Investigate the Efficacy, Safety and Tolerability of AZD1152 Alone and in Combination With Low Dose Cytosine Arabinoside (LDAC)in Acute Myeloid Leukaemia (AML) Patients
Acronym: SPARK-AML1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1531C00009
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukaemia,; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — 2-((3-((4-((5-(2-((3-fluorophenyl)amino)-2-oxoethyl)-1H-pyrazol-3-yl)amino)quinazolin-7-yl)oxy)propyl)(ethyl)amino)ethyl dihydrogen phosphate

ARMS (2):
- AZD1152 1200 mg (Experimental): AZD1152 1200 mg, iv, 7 day infusion monotherapy
  Interventions: Drug: AZD1152
- LDAC 20 mg (Active Comparator): LDAC 20 mg, sc, bd, 10 days (400mg per cycle)
  Interventions: Drug: LDAC

INTERVENTIONS:
Drug: AZD1152 — 1200 mg, iv, 7 day infusion
  Arms: AZD1152 1200 mg
Drug: LDAC — 20 mg, sc, bd, 10 days
  Arms: LDAC 20 mg

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of AZD1152 alone and in combination with low dose cytosine arabinoside (LDAC) in comparison with LDAC alone in AML patients.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Newly diagnosed male or female patients aged 60 and over
* De Novo or Secondary AML
* Not eligible for intensive induction with anthracycline-based combination chemotherapy as a result of at least one of the following:Age ≥75 years; Adverse cytogenetics, e.g., as defined by the MRC Prognostic Groupings; WHO performance status >2; Organ dysfunction arising from significant co-morbidities not directly linked to leukaemia

Exclusion Criteria:

* Participation in another clinical study in which an investigational product was received within 14 days before the first dose in this study, or at any time if the patient has not recovered from side-effects associated with that investigational product
* Administration of LDAC is clinically contraindicated
* Patients with AML of FAB M3 classification Acute Promyelocytic Leukaemia (APL)
* Patients with blast crisis of chronic myeloid leukaemia

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Stockman, Study Director — AstraZeneca; Hagop Kantarjian, Principal Investigator — M.D. Anderson Cancer Center
Locations (45):
- United States (8):
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Greenville, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
- Australia (4):
  - Research Site, Westmead, New South Wales
  - Research Site, Herston, Queensland
  - Research Site, Melbourne, Victoria
  - Research Site, Parkville, Victoria
- France (6):
  - Research Site, Angers
  - Research Site, Clermont-Ferrand
  - Research Site, Grenoble
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Nantes
- Germany (5):
  - Research Site, Duisburg
  - Research Site, Erlangen
  - Research Site, Frankfurt
  - Research Site, Münster
  - Research Site, Villingen-Schwenningen
- Italy (5):
  - Research Site, Bologna, BO
  - Research Site, Genova, GE
  - Research Site, Orbassano, TO
  - Research Site, Udine, UD
  - Research Site, Roma
- Japan (7):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Yoshida-gun, Fukui
  - Research Site, Maebashi, Gunma
  - Research Site, Isehara, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Chūō, Tokyo
  - Research Site, Fukuoka
- Romania (2):
  - Research Site, Brasov
  - Research Site, TG Mures
- Spain (6):
  - Research Site, Badalona(barcelona), Catalonia
  - Research Site, Barcelona, Catalonia
  - Research Site, Madrid, Madrid
  - Research Site, Majadahonda, Madrid
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Valencia, Valencia
- United Kingdom (2):
  - Research Site, Brighton
  - Research Site, London

REFERENCES:
- [Derived] Quintas-Cardama A, Ravandi F, Liu-Dumlao T, Brandt M, Faderl S, Pierce S, Borthakur G, Garcia-Manero G, Cortes J, Kantarjian H. Epigenetic therapy is associated with similar survival compared with intensive chemotherapy in older patients with newly diagnosed acute myeloid leukemia. Blood. 2012 Dec 6;120(24):4840-5. doi: 10.1182/blood-2012-06-436055. Epub 2012 Oct 15. PMID 23071272

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient was randomized on 22/07/2009 and last patient last visit has occurred on 27/06/2011.
Groups:
- AZD1152 1200mg: AZD1152 1200 mg, iv, 7 day infusion monotherapy
- LDAC 20mg: LDAC 20 mg, sc, bd, 10 days (400mg per cycle)
Period: Overall Study
Arm/Group | AZD1152 1200mg | LDAC 20mg
Started | 48 | 26
Completed | 12 | 2
Not Completed | 36 | 24
Not completed — Death | 28 | 13
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Lack of Efficacy | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1152 1200mg | LDAC 20mg | Total
Number analyzed (Participants) | 48 | 26 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.3 (5.79) | 71.5 (5.75) | 74.0 (6.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 8 | 31
  Male | 25 | 18 | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Overall Complete Response for Stage I
Description: Percentage of patients achieving either a complete response (CR) or a confirmed complete remission with incomplete recovery of neutrophils or platelets (confirmed CRi). Per Cheson Criteria: Confirmed complete remission (CRi) is defined as a disappearance of blasts in the peripheral blood; a decrease in bone marrow blasts to <5% total bone marrow nucleated cells demonstrated in bone marrow aspirate; absence of Auer rods; no persistent extramedullary leukaemia. Complete response (CR) is defined as all requirements to meet CRi and in addition: recovery of neutrophils to ≥1.0 x 109/L and platelets to ≥100 x 109/L; transfusion-independence.
Time Frame: IWG Cheson criteria every 28 days from randomization for study duration (24 months, between 2009 - 2011)
Population: modified Intent to Treat (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | AZD1152 1200mg | LDAC 20mg
Number analyzed (Participants) | 48 | 26
percentage of participants | 35.4 | 11.5

2. Secondary Outcome: Duration of Response (DoR): Stage I and Transition Phase
Description: DoR was defined for the median of days which showed a confirmed CRi or CR, as the time from first documented evidence of CRi or CR until the first documented sign of disease progression or death. Duration of Response was measured from the Response Start date until evidence of patient relapse or death. Stage I : 45 patients randomized in a 2:1 ratio to AZD1152 or LDAC. Transition phase: enrollment of up to 30 additional patients randomized as per stage I.
Time Frame: DoR was measured every 28 days from randomization for study duration (24 months, between 2009 - 2011)
Population: modified Intent to Treat (mITT)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | AZD1152 1200mg | LDAC 20mg
Number analyzed (Participants) | 17 | 3
days | 82 [43 to 189] | NA [NA to NA] — This was not calculable because there were only 3 responses (events) in this group and the method of estimating the median was using Kaplan-Meier methods.

3. Secondary Outcome: Disease Free Survival (DFS)
Description: Disease-free Survival is defined as the time from randomisation to relapse or death from any cause.
Time Frame: DFS was measured every 28 days from randomization for study duration (24 months, between 2009 - 2011)
Population: modified Intent to Treat (mITT)
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | AZD1152 1200mg | LDAC 20mg
Number analyzed (Participants) | 17 | 3
months | 5.6 [3.3 to 7.9] | NA [NA to NA] — This was not calculable because there were only 3 responses (events) in this group and the method of estimating the median was using Kaplan-Meier methods.

4. Secondary Outcome: Time To Complete Response (TTCR)
Description: TTCR is measured as time from randomization to either a complete response (CR) or a confirmed complete remission with incomplete recovery of neutrophils or platelets (confirmed CRi)
Time Frame: Response was measured every 28 days from randomization for study duration (24 months, between 2009 - 2011)
Population: modified Intent to Treat (mITT)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | AZD1152 1200mg | LDAC 20mg
Number analyzed (Participants) | 17 | 3
days | 59 [27 to 180] | 64 [63 to 96]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is defined as the median time from randomisation to death from any cause. Patients who were not known to have died at the time of the analysis were censored at the date they were last known to be alive.
Time Frame: Assessed from randomisation until the date of death from any cause, assessed up to 24 months
Population: modified Intent to Treat (mITT)
Measure: Median (Full Range); unit: months
Arm/Group | AZD1152 1200mg | LDAC 20mg
Number analyzed (Participants) | 48 | 26
months | 8.2 (43) [0.1 to 15.9] | 4.5 (32) [0.2 to 20.4]

6. Secondary Outcome: Percent of Patients With Worsened Trial Outcome Index (TOI)
Description: TOI is derived from the sum of the Functional Well Being (FWB), Physical Well Being (PWB) and additional subscales of the FACT-Leu. The TOI subscale consists of 31 items with TOI scores ranging from 0 to 124. The TOI is described as a summary measure of HRQoL. Higher scores indicate better HRQoL. Negative changes from baseline indicate a worsening of HRQoL while positive changes indicate an improvement in HRQoL. A response of "Worsened" was a change from baseline in score of less than or equal to -9.
Time Frame: TOI was measured every 28 days from randomization for study duration (24 months, between 2009 - 2011)
Population: modified Intent to Treat (mITT)
Measure: Number; unit: percentage of participants
Arm/Group | AZD1152 1200mg | LDAC 20mg
Number analyzed (Participants) | 48 | 26
percentage of participants | 31.3 | 11.5

7. Secondary Outcome: Percent of Patients With Worsened Functional Assessment of Cancer Therapy - Leukaemia (FACT-Leu) Score.
Description: The total FACT-Leu score consists of 44 items with total scores ranging from 0 to 176. Higher scores indicate better HRQoL. Negative changes from baseline indicate a worsening of HRQoL while positive changes indicate an improvement in HRQoL. A response of "Worsened" was a change from baseline in score of less than or equal to -11.
Time Frame: FACT-Leu was measured every 28 days from randomization for study duration (24 months, between 2009 - 2011)
Population: modified Intent to Treat (mITT)
Measure: Number; unit: percentage of participants
Arm/Group | AZD1152 1200mg | LDAC 20mg
Number analyzed (Participants) | 48 | 26
percentage of participants | 29.2 | 11.5

ADVERSE EVENTS:
Arm/Group | AZD1152 1200mg | LDAC 20mg
Serious Adverse Events (participants affected / at risk) | 23/48 | 10/26
Other Adverse Events (participants affected / at risk) | 33/48 | 10/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1152 1200mg (N=48) | LDAC 20mg (N=26)
Febrile Neutropenia (Blood and lymphatic system disorders) | 5 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile Bone Marrow Aplasia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Myocardial Ischaemia (Cardiac disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 0
Pyrexia (General disorders) | 4 | 1
Device Occlusion (General disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 2
Arthritis Infective (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium Difficile Sepsis (Infections and infestations) | 0 | 1
Enterococcal Bacteraemia (Infections and infestations) | 1 | 0
Escherichia Infection (Infections and infestations) | 1 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 0 | 1
Neutropenic Sepsis (Infections and infestations) | 0 | 1
Oral Candidiasis (Infections and infestations) | 1 | 0
Pulmonary Mycosis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0
White Blood Cell Count Increased (Investigations) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Blast Cell Proliferation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1152 1200mg (N=48) | LDAC 20mg (N=26)
Febrile Neutropenia (Blood and lymphatic system disorders) | 32 | 5
Anaemia (Blood and lymphatic system disorders) | 12 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 6
Leukopenia (Blood and lymphatic system disorders) | 6 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 2
Lymphopenia (Blood and lymphatic system disorders) | 4 | 0
Coagulopathy (Blood and lymphatic system disorders) | 3 | 1
Tachycardia (Cardiac disorders) | 3 | 3
Vertigo (Ear and labyrinth disorders) | 3 | 0
Conjunctival Haemorrhage (Eye disorders) | 3 | 0
Stomatitis (Gastrointestinal disorders) | 33 | 4
Diarrhoea (Gastrointestinal disorders) | 24 | 3
Constipation (Gastrointestinal disorders) | 23 | 8
Nausea (Gastrointestinal disorders) | 21 | 10
Vomiting (Gastrointestinal disorders) | 17 | 5
Haemorrhoids (Gastrointestinal disorders) | 7 | 1
Oral Pain (Gastrointestinal disorders) | 5 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 4
Dry Mouth (Gastrointestinal disorders) | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 0
Dysphagia (Gastrointestinal disorders) | 4 | 1
Tongue Ulceration (Gastrointestinal disorders) | 4 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 0
Gingival Bleeding (Gastrointestinal disorders) | 3 | 3
Toothache (Gastrointestinal disorders) | 3 | 0
Pyrexia (General disorders) | 13 | 8
Fatigue (General disorders) | 9 | 6
Asthenia (General disorders) | 7 | 8
Oedema Peripheral (General disorders) | 8 | 7
Hyperthermia (General disorders) | 5 | 0
Oedema (General disorders) | 4 | 1
Pain (General disorders) | 4 | 1
Catheter Site Pain (General disorders) | 3 | 2
Catheter Site Related Reaction (General disorders) | 3 | 0
Chills (General disorders) | 3 | 3
Catheter Site Haematoma (General disorders) | 0 | 2
Injection Site Haematoma (General disorders) | 0 | 2
Pneumonia (Infections and infestations) | 6 | 1
Sepsis (Infections and infestations) | 6 | 0
Oral Candidiasis (Infections and infestations) | 5 | 0
Bacteraemia (Infections and infestations) | 3 | 0
Cellulitis (Infections and infestations) | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 1
Alanine Aminotransferase Increased (Investigations) | 4 | 0
Weight Decreased (Investigations) | 3 | 4
Blood Creatinine Increased (Investigations) | 3 | 1
Breath Sounds Abnormal (Investigations) | 3 | 0
Blood Pressure Decreased (Investigations) | 0 | 2
Weight Increased (Investigations) | 0 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 10 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 8 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Joint Swelling (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 8 | 1
Dysgeusia (Nervous system disorders) | 5 | 0
Dizziness (Nervous system disorders) | 4 | 4
Insomnia (Psychiatric disorders) | 11 | 3
Anxiety (Psychiatric disorders) | 4 | 1
Confusional State (Psychiatric disorders) | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 0
Rash (Skin and subcutaneous tissue disorders) | 10 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 4
Petechiae (Skin and subcutaneous tissue disorders) | 4 | 4
Erythema (Skin and subcutaneous tissue disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 2
Hypotension (Vascular disorders) | 5 | 1
Haematoma (Vascular disorders) | 2 | 3
Pallor (Vascular disorders) | 0 | 2
Phlebitis (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less